CLINICAL TRIAL: NCT04849234
Title: FirstCRY Study : Acoustic Analysis of the First Babies Crying in Delivery Room and Adaptation to Extra Uterine Life
Brief Title: Acoustic Analysis of the First Babies Crying in Delivery Room and Adaptation to Extra Uterine Life
Acronym: FIRSTCRY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN262021/CHUSTE
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Premature Birth
Keywords: Crying; Apgar score; Infant Behavior; First cry; delivery room; extra uterine life
MeSH Terms: conditions — Premature Birth; Crying; Infant Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New born: New born population aged 37 Weeks of Amenorrhea (SA) to 42 Weeks of Amenorrhea (SA) will be included. Their cries will be longitudinally registered.
  Interventions: Behavioral: newborn cries

INTERVENTIONS:
Behavioral: newborn cries — Their cries will be longitudinally registered from the age of birth until the first 15 minutes of birth using an automatic record device: Recorder ZOOM H4N.
  The wav-sized files obtained from each recording will then be analyzed indiscriminately via an acoustic processing script created for the PRAAT software® by the post-doctoral fellows of the ENES laboratory (Sensory NeuroEthology Team) on the site of the Faculty of Sciences of Saint-Etienne.

SUMMARY:
Interpreting the cry of new-borns is a real challenge not only for perinatal professionals but also for parents, who are confronted daily with those sounds.

The description and the acoustic analysis of baby's cry can allow healthcare professionals to better adapt their care during the first months of life.

Thanks to an objective analysis method as acoustic analysis, the particularities of the first cry should provide us information on the quality of adaptation to ambient air life.

DETAILED DESCRIPTION:
Interpreting the cry of new-borns is a real challenge not only for perinatal professionals but also for parents, who are confronted daily with those sounds.

The description and the acoustic analysis of baby's cry can allow healthcare professionals to better adapt their care during the first months of life. Aiming for this objective, many studies have already been carried out on infants crying in the first months of life, in order to better understand their significance (pain, discomfort, hunger) and the mechanisms of recognition and discrimination by parents or listeners. Various techniques are promising to characterize the acoustic space of cry (maximum frequency, intensity, harmonics, duration…).

However, few studies have investigated the acoustic characteristics of the first cry of life in the delivery room. Its intensity and characteristics are closely related to the laryngeal anatomy and respiratory capacity. Thus, a vigorous cry with its own acoustic characteristics could be the witness of a good adaptation to extra uterine life, while a weak or plaintive cry should warn the caregiver on difficulties in this adaptation.

Thanks to an objective analysis method as acoustic analysis, the particularities of the first cry should provide us information on the quality of adaptation to ambient air life.

The investigators hypothesize that the acoustic characteristics of the first cries of newborns recorded at birth are correlated with the criteria of extra uterine life adaptation (Apgar score, pH and lactates collected from the umbilical cord), with the respiratory score (Silverman) and with the early neonatal outcome (transfer to the intensive care unit).

ELIGIBILITY:
Inclusion Criteria:

* Infant born between 37 and 42 SA
* Live infant at birth
* Parent who received informed written information about the study

Exclusion Criteria:

- Emergency after childbirth (haemorrhage)

Ages: 1 Minute to 15 Minutes | Sex: All
Age Groups: Child
Study Population: Infant newborn
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-02 (Actual)

PRIMARY OUTCOMES:
Fo : maximum fundamental frequency (Hz) of the cry | During the first 15 minutes of life
  Measured by device: Recorder ZOOM H4N and analyzed with PRAAT® software
  The F0 and Apgar score will be correlated
Apgar score (0-10) | During the first 15 minutes of life
  The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting score ranges from zero to 10.
  The five criteria are : appearance, pulse, grimace, activity, respiration.
  The F0 and Apgar score will be correlated

SECONDARY OUTCOMES:
Pitch of the cry (Hz) Crying acoustic structures | During the first 15 minutes of life
  Measured by device: Recorder ZOOM H4N and analyzed with PRAAT® software
roughness of the cry (Hz) | During the first 15 minutes of life
  Measured by device: Recorder ZOOM H4N and analyzed with PRAAT® software
Duration of cry (s) | During the first 15 minutes of life
  Measured by device: Recorder ZOOM H4N and analyzed with PRAAT® software
Number of cry | During the first 15 minutes of life
  Measured by device: Recorder ZOOM H4N and analyzed with PRAAT® software

CONTACTS AND LOCATIONS:
Overall Officials: HUGUES PATURAL, MD PHD, Principal Investigator — CHU ST ETIENNE FRANCE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No